CLINICAL TRIAL: NCT04326127
Title: Performance Evaluation of the Compumedics "Somfit" Sleep Monitoring Device
Brief Title: Evaluation of Compumedics "Somfit" Device
Status: Completed | Type: Observational
Sponsor: Compumedics Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: SOMFIT02
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Healthy volunteers
  Interventions: Device: Intervention is the validation of a sleep monitoring device (i.e. Somfit) against the gold-standard polysomnograph with electroencephalograph (i.e. the Greal system)
- Case: Volunteers with diagnosed sleep apnea
  Interventions: Device: Intervention is the validation of a sleep monitoring device (i.e. Somfit) against the gold-standard polysomnograph with electroencephalograph (i.e. the Greal system)

INTERVENTIONS:
Device: Intervention is the validation of a sleep monitoring device (i.e. Somfit) against the gold-standard polysomnograph with electroencephalograph (i.e. the Greal system) — Data were recorded overnight by both devices simultaneously

SUMMARY:
To study whether Somfit is substantially equivalent to an existing approved device (i.e. Compumedic's Grael System) to assist in elucidating sleep disorders.

DETAILED DESCRIPTION:
Sleep is recognized as one of the three pillars of health (i.e. nutrition, exercise and sleep). Poor quality and fragmented sleep leads to an increase in the risk for development of chronic health conditions. Given the importance of good quality sleep and its critical role in overall well-being, there is a need for regular monitoring and assessment of sleep quality in individuals. However, current technologies will only allow for this to be performed in sleep clinics and with the help of full polysomnography (PSG) systems which require the patients to spend a night at the clinic with several wired electrodes connected to their scalp. This will cause discomfort for the patients in a long run. To solve this problem, Compumedics has recently developed a miniaturized, portable and affordable sleep monitoring system with code name of "Somfit" which can be used in the comfort of patients' home. The aim of this study is to validate Somfit for home based sleep studies.

ELIGIBILITY:
Inclusion Criteria:

* Individuals age between 18 to 75
* Be able to give informed consent
* Individuals with diagnosed Obstructive Sleep Apnoea (OSA)

Exclusion Criteria:

* Less than 18 years of age
* Greater than 75 years of age
* Unable or not willing to provide informed consent
* Need for nursing care
* Currently working nightshift

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 volunteers were invited to participate in this study. 15 participants will be selected among healthy volunteers, by advertising to the general public. The remaining 15 will be among patients with diagnosed sleep apnea who visit SleepMetrics clinic as part of their routine treatment.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Comparison between raw EEG signals | single night recording for each subject
  Direct comparison of Raw EEG data between Somfit and Grael system on an epoch by epoch basis (with each epoch being equivalent to 30 secs) to test and validate Somfit for data acquisition, display and record of Raw EEG data.

SECONDARY OUTCOMES:
Comparison between Manual and Automatic sleep Scoring - Sleep hypnogram | single night recording for each subject
  Epoch-by-epoch comparison between manual and automatic scoring of sleep data recorded by Somfit and Grael devices

OTHER OUTCOMES:
Validation of the new device for detection of sleep apnea | single night recording for each subject
  Differentiation between case and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Kealy, Principal Investigator — Sleepmetrics
Locations (1):
- SleepMetrics Pty Ltd, Melbourne, Victoria, Australia